CLINICAL TRIAL: NCT00974324
Title: Phase 2 Study of Endostar Combined With CHOP Regimen as the First Line Chemotherapy for Untreated Peripheral T Cell Lymphoma
Brief Title: Endostar Combined With CHOP Regimen as First Line Chemotherapy for Peripheral T Cell Lymphoma
Acronym: PTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Haiyi Guo, Medical Oncology of Fudan University Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL0908
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: T Cell Lymphoma
Keywords: peripheral T cell lymphoma; chemotherapy; anti-angiogeneses
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, T-Cell, Peripheral | interventions — endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): endostar combined with CHOP regimen
  Interventions: Drug: endostar and CHOP

INTERVENTIONS:
Drug: endostar and CHOP — endostar, 7.5m g/m2, intravenous, Day 2-15, repeat every 3 weeks
  CHOP: Cyclophosphamide, Hydroxydaunorubicin, Oncovin, Prednisone
  Other Names: endostar

SUMMARY:
The role of angiogenesis has been less clear in lymphoma than in solid tumors, in part related to the heterogeneity of disease and technical issues. In addition to vascular endothelial growth factor (VEGF) effects on angiogenesis and the integrity of tumor vasculature, autocrine VEGF-receptor (VEGF-R)-mediated signaling may play a role in lymphoma. Microvessel density, a measure of angiogenesis, is highest in peripheral T-cell lymphomas (PTCL), followed by diffuse large B-cell (DLBCL) and intra-follicular follicular lymphoma (FL).

DETAILED DESCRIPTION:
To investigate efficacy and safety of endostar combined with CHOP regimen as first line treatment for peripheral T cell lymphoma.The second subject is to clarify the association between expression of VEGF and prognosis in peripheral T cell lymphoma,unspecified(PTCL-U) and angioimmunoblastic T-cellLymphoma(AILT).Methods 15 cases of PTCL were enrolled in this study.Immunohistochemical staining was performed by EnVision method using antibodies VEGF.

ELIGIBILITY:
Inclusion Criteria:

* Disease Characteristics:

  * Diagnosis of peripheral T-cell:

    * Any stage disease allowed
  * At least 1 objective measurable disease parameter
  * No anaplastic lymphoma kinase (ALK)-positive T-cell large cell lymphoma

    * ALK-negative T-cell large cell lymphoma allowed
  * No cutaneous T-cell lymphoma

    * No sezary syndrome
    * No NK/T cell lymphoma
  * No history of or current radiographic evidence of CNS metastasis, including previously treated, resected, or asymptomatic brain lesions or leptomeningeal involvement
* Patient Characteristics:

  * Age:

    * 18 -75 years
  * Performance status:

    * ECOG 0-2
  * Life expectancy:

    * No less than 12 weeks
  * Hematopoietic:

    * Absolute neutrophil count ≥ 1,500/mm^3
    * Hemoglobulin ≥ 80*10^12/L
    * Platelet count ≥ 100,000/mm^3
    * No evidence of bleeding diathesis or coagulopathy
  * Hepatic:

    * Bilirubin ≤ 1.5 mg/dL
    * AST ≤ 2.5 times ULN
    * PT, INR, and PTT ≤ 1.5 times normal
  * Renal:

    * Creatinine ≤ 1.5 times normal
  * Cardiovascular:

    * No cerebrovascular accident within the past 6 months
    * No myocardial infarction within the past 6 months
    * No unstable angina within the past 6 months
    * No New York Heart Association class II-IV congestive heart failure
    * No uncontrolled hypertension (i.e., systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 100 mm Hg)
    * No other clinically significant cardiovascular or peripheral vascular disease
    * LVEF is normal
  * Other:

    * Not pregnant or nursing
    * Fertile patients must use effective contraception
    * No history of active seizures
    * No non-healing ulcer (unless involved with lymphoma)
    * No active infection requiring parenteral antibiotics
    * No known HIV positivity
    * No other active malignancy within the past 6 months except carcinoma in situ of the cervix or basal cell carcinoma of the skin
* PRIOR CONCURRENT THERAPY:

  * Biologic therapy:

    * Not specified
  * Chemotherapy:

    * No prior chemotherapy was allowed
  * Surgery:

    * More than 4 weeks since prior major invasive surgery or open biopsy
    * At least 7 days since prior minor surgery
    * No concurrent major surgery

Exclusion Criteria:

* Prior treatment included chemotherapy and radiotherapy
* With the following risk factors: Uncontrolled or severe cardiovascular disease (e.g., myocardial infarction within the past 6 months, congestive heart failure treated with medications, or uncontrolled hypertension)
* Pregnant or nursing
* Other currently active malignancy except nonmelanoma skin cancer
* Uncontrolled or severe bleeding,diarrhea,intestinal obstruction
* Hypersensitivity to albumen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
efficacy include overall response rate, disease free survival and overall survival | 1 year

SECONDARY OUTCOMES:
safety of endostar combined with CHOP | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Junning Cao, MD, Principal Investigator — Member of Fudan University Cancer Hospital
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China